CLINICAL TRIAL: NCT01997619
Title: Biological Mesh Repair of Complex Ventral Hernias in High Risk Patients
Brief Title: Biological Mesh Repair of Complex Hernias in High Risk Patients
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Louise Preisler, MD, Rigshospitalet, Denmark
Other Study IDs: 30245705
Record Dates: First submitted 2013-11-24; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Hernia
Keywords: biological mesh; contaminated hernia; abdominal wall reconstruction
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Complex ventral hernia repair is a significant surgical challenge with high frequencies of both wound complications and recurrence. The Ventral Hernia Working Group (VHWG) described in 2010 recommendations regarding grading and technique of repair, which we have followed since November 2011.The purpose of the this study was to evaluate our results after biologic mesh repair of complex hernias.

DETAILED DESCRIPTION:
Obervational study

Primare outcome: Surgical site occurence

Secondary outcome: Hernia recurrence

Biolocal mesh: Ventral hernia repair in a population with severe co-morbidity and contaminated hernia.

ELIGIBILITY:
Inclusion Criteria: Abdominal wall reconstruction with biological mesh -

Exclusion Criteria: Pregancy,

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 16 consecutive patients with biological mesh repair
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
surgical site occurence | 30 days
  Wound infections, redness, seromas, dehiesience at the hernia implant site

SECONDARY OUTCOMES:
hernia recurrence | 20 months
  Hernia recurrence at the hernia implant site

CONTACTS AND LOCATIONS:
Overall Officials: Linda Bardram, MD, Study Chair — Rigshospitalet, Copenhagen, University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen, Denmark